CLINICAL TRIAL: NCT01054378
Title: Diaphragmatic Movement Before and After Stellate Ganglion Block : A Ultrasonographic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Duck Mi Yoon/Professor of Anesthesiology and Pain Medicine,, Yonsei University College of Medicine, Seoul, South Korea,
Purpose: Treatment
Other Study IDs: 4-2009-0614
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Head Pain; Neck Pain; Shoulder Pain; Arm Pain; Neural Sensory Hearing Loss
MeSH Terms: conditions — Headache; Neck Pain; Shoulder Pain

INTERVENTIONS:
Procedure: M-mode ultrasonography — Evaluation of diaphragmatic movement using M-mode ultrasonography before and after stellate ganglion block with 1% lidocaine

SUMMARY:
The temporary diaphrgmatic dysfunction will occur after stellate ganglion block(SGB) and will be easily detected by M-mode ultrasonography

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II patients who have head and neck pain or shoulder pain or sudden sensory neural hearing loss

Exclusion Criteria:

* coagulopathy, pulmonary disease, neuropathy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The amplitude of diaphragm movement before and after SGB during quiet breathing, deep breathing and voluntary sniff, inspiratory time and expiratory time, oxygen saturation | The ultrasonographic evaluation will take place just before and 30 minutes after stellate ganglion block.

CONTACTS AND LOCATIONS:
Overall Officials: Duck Mi Yoon, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea